CLINICAL TRIAL: NCT01834040
Title: Study Safety and Efficacy of of AUTOLOGOUS Bone Marrow Derived Mono Nuclear Stem Cell (BMMNCs) for the Patient With Duchenne Muscular Dystrophy. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Study Safety and Efficacy of BMMNC for the Patient With Duchenne Muscular Dystrophy
Acronym: BMMNC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00102
Record Dates: First submitted 2013-02-26; First posted 2013-04-17 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Muscular Dystrophy; Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; Muscular Dystrophy; Myopathy
MeSH Terms: conditions — Muscular Dystrophies; Muscular Dystrophy, Duchenne; Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intralesional and Intravenous (Other): Intralesional/ Intravenous of Autologous Stem cells.
  Interventions: Other: Intralesional/ Intravenous of Autologous Stem cells.

INTERVENTIONS:
Other: Intralesional/ Intravenous of Autologous Stem cells. — Intralesional/ Intravenous of Autologous MNCs per dose
  Other Names: Intralesional/ Intravenous of Autologous MNCs.; Intralesional/ Intravenous of Autologous MNCs

SUMMARY:
This Study is single arm, single center trial to check the safety and efficacy of BMMNC (100 million per dose) for the patient with Duchenne Muscular Dystrophy,

DETAILED DESCRIPTION:
Muscular dystrophies, or MD, are a group of inherited conditions, which means they are passed down through families. They may occur in childhood or adulthood. There are many different types of muscular dystrophy. They include:

Duchenne muscular dystrophy is a form of muscular dystrophy that worsens quickly. Other muscular dystrophy (including Becker's muscular dystrophy) get worse much more slowly.

Duchenne muscular dystrophy is caused by a defective gene for dystrophin (a protein in the muscles). However, it often occurs in people without a known family history of the condition.

Symptoms usually appear before age 6 and may appear as early as infancy. They may include:

Fatigue

Learning difficulties (the IQ (intelligence quotient )can be below 75)

Intellectual disability (possible, but does not get worse over time)

Muscle weakness

Begins in the legs and pelvis, but also occurs less severely in the arms, neck, and other areas of the body

Difficulty with motor skills (running, hopping, jumping)

Frequent falls

Trouble getting up from a lying position or climbing stairs

Weakness quickly gets worse

Progressive difficulty walking

Ability to walk may be lost by age 12, and the child will have to use a wheelchair

Breathing difficulties and heart disease usually start by age 20

ELIGIBILITY:
Inclusion Criteria:

* Patient with Diagnose of Duchenne Muscular Dystrophy.
* Aged in between 4 to 20 Years.
* Willingness to undergo Bone Marrow derived Autologous cell Therapy.
* Ability to comprehend the explained protocol and thereafter give an informed consent as well as sign the required Informed Consent form(ICF) for the study.
* Ability and willingness to regular visit to hospital for protocol procedures and follow up

Exclusion Criteria:

* Patient with History of Immunodeficiency HIV+,Hepatitis B ,HBV and TPPA+, Tumor Markers+
* Patients with History of Hypertension and Hypersensitive.
* Patient who is not Diagnose of Duchenne Muscular Dystrophy.
* Alcohol and drug abuse / dependence.

Ages: 4 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Improvement of daily living scale. | 6 MONTH

SECONDARY OUTCOMES:
Improvement of Muscular dystrophy specific functional Rating scale | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India